CLINICAL TRIAL: NCT00929682
Title: Levobupivacaine for Epidural Analgesia in Labour
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: CHU-0055
Record Dates: First submitted 2009-06-26; First posted 2009-06-29 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Analgesia, Epidural
Keywords: Labor; Epidural analgesia; Local anesthetics; Levobupivacaine; Opiates; Patient-controlled; Active spontaneous labor requiring epidural analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Levobupivacaine 0.568mg.mL (Experimental)
  Interventions: Drug: Randomization between two referenced treatments
- Levobupivacaine 1.136mg.mL (Other)
  Interventions: Drug: Randomization between two referenced treatments

INTERVENTIONS:
Drug: Randomization between two referenced treatments — Levobupivacaine 0.568 mg.mL-1 and sufentanil 0.45 g.mL-1, 20 mL epidurally for induction, then by a patient-controlled regimen with 5-mL self-administered boli in addition to a continuous infusion of 5 mL.hr-1.
  Same protocol, with levobupivacaine 1.136 mg.mL-1 and sufentanil 0.45 g.mL-1.

SUMMARY:
In a prospective randomised study involving primiparous women in spontaneous uncomplicated labour with cervical dilatation > 7 cm, epidural analgesia will be given with an initial volume of 20 mL anaesthetic solution, followed by a standardised algorithm of top-up manual injections to achieve analgesia, then by a patient-controlled regimen with 5-mL self-administered boli in addition to a continuous infusion of 5 mL.hr-1. The anaesthetic solution will be levobupivacaine presented in 100-mL bags from the market, 0.0625%, or 0.125%, in which 10 mL (50 µg) of sufentanil will be added. The final concentrations will be 0.568 and 1.136 mg.mL-1 respectively, both with sufentanil 0.45 µg.mL-1. Parturients and midwifes assessing pain during labour will be blinded to the design

DETAILED DESCRIPTION:
Since epidural analgesia has been developed to relieve labour pain, many solutions have emerged to lower risk / efficacy ratio, by using low-concentrated and/or less toxic local anaesthetics. Levobupicaine emerges as a safer alternative than its racemic parent . It is available on the French market in pre-filled bags with two different concentrations (0.625 and 1.25 mg.mL-1), both indicated for analgesia in postoperative context and in labour, without more precision. Presentation in bags allows preparing once at the initiation of epidural analgesia a solution usable throughout labour, leading the anaesthetist to a univocal choice, mostly following his/her personal beliefs. Our aim is to compare the effects of epidural analgesia under these two presentations. Sufentanil will be added to levobupicaine whatever the concentration used. This trial is conducted in primiparous, in which pain during labour is commonly more resistant to relief.

ELIGIBILITY:
Inclusion Criteria:

* Parturient > 18 years old
* ASA physical status 1 or 2
* Primiparity
* Singleton
* Gestational age > 36 weeks
* Spontaneous labour with cervical dilatation > 7 cm

Exclusion Criteria:

* Gestational age < 36 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2007-06; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
- Spontaneous pain during labour (on VAS). - Number of required additional epidural boluses, either self-administered or medically given as a rescue. | during labour

SECONDARY OUTCOMES:
- Pain at delivery - Pain at post-delivery sutures - Motor block - Duration of labour - Obstetrical events (cesarean, instrumental delivery) | during labour

CONTACTS AND LOCATIONS:
Overall Officials: Martine Bonnin, MB, Principal Investigator — University Hospital, Clermont-Ferrand

REFERENCES:
- [Result] Tixier S, Bonnin M, Bolandard F, Vernis L, Lavergne B, Bazin JE, Duale C. Continuous patient-controlled epidural infusion of levobupivacaine plus sufentanil in labouring primiparous women: effects of concentration. Anaesthesia. 2010 Jun;65(6):573-580. doi: 10.1111/j.1365-2044.2010.06369.x. PMID 20565392
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/20565392